CLINICAL TRIAL: NCT04730882
Title: Effect of Postprandial Hyperglycemia on Vasculature in Type 1 Diabetes and Healthy Adults
Acronym: WBH001
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, William Horton, MD, Principal Investigator, University of Virginia
Other Study IDs: 200216; KL2TR003016 (NIH)
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes; Hyperglycemia, Postprandial
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Control: Healthy subjects 18-35 years of age
  Interventions: Dietary Supplement: Mixed Meal
- Type 1 Diabetes: People with type 1 diabetes (18-35 yrs) who have type 1 diabetes based on WHO diagnostic criteria for > 1 year
  Interventions: Dietary Supplement: Mixed Meal

INTERVENTIONS:
Dietary Supplement: Mixed Meal — the meal will be 40% of each subject's daily estimated caloric need, with 50%, 30%, 20% from carbohydrates, fat and protein, respectively

SUMMARY:
To the investigator's knowledge, there are no data available in the current literature regarding the acute effects of postprandial hyperglycemia and insulin timing on myocardial perfusion in people with type 1 diabetes (T1D). Observational studies using CEU in type 2 diabetes demonstrate that postprandial hyperglycemia determines myocardial perfusion defects. The investigator hypothesizes that the combination of postprandial hyperglycemia and insulin increases pulse wave velocity (i.e., aortic stiffness) and myocardial vasoconstriction, thereby reducing myocardial perfusion in T1D when compared to healthy controls. Furthermore, the investigator hypothesizes in T1D that dosing insulin before meal intake will ameliorate these cardiovascular defects.

DETAILED DESCRIPTION:
The investigator will compare 17 T1D and 17 age-, sex-, and BMI-matched healthy controls (18-35 yrs) measuring pulse wave velocity (PWV), flow-mediated dilation (FMD) and myocardial perfusion (contrast enhanced ultrasound [CEU]) before and 2 hours after ingesting a mixed meal (40% of each subject's daily estimated caloric need, with 50%, 30%, 20% from carbohydrates, fat and protein, respectively).

T1D participants will have 2 study admissions:

A) injection of insulin 15 minutes before ingesting a mixed meal. B) injection of insulin 15 min after ingesting a mixed meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy with no chronic illness

  * Age 18-35 years
  * BMI ≤ 30 (wt kg/ht m2)
  * Normal screening labs or no clinically significant values
  * T1D participants must have T1D based on WHO diagnostic criteria for > 1 year

    * A fasting plasma glucose level >126 mg/dl (7.0 mmol/l)
    * A casual plasma glucose >200 mg/dl (11.1 mmol/l)
    * In the absence of unequivocal hyperglycemia, the diagnosis must be confirmed on a subsequent day.
  * Subjects using sensor-augmented insulin pump therapy and/or artificial pancreas (closed loop system) will be included

Exclusion Criteria:

* • Smoking presently or have quit < 2 years.

  * BP >140/90 mmHg
  * BMI >30 (wt kg/ht m2)
  * Pulse oximetry <90%
  * Elevated LDL cholesterol > 160 mg/dl
  * HbA1c ≥ 9 %
  * Use of statins, calcium channel blocker, ACE, ARB, nitrates, alpha-beta blockers or diuretics
  * History of cardiac, cerebrovascular, gastrointestinal, liver, renal decease or cancer
  * Presence of an intracardiac or intrapulmonary shunt (we will screen for this by auscultation during the physical exam by PI).
  * Retinopathy (beyond mild non proliferative retinopathy)
  * Urine albumin/creatinine ratio > 300 mg per g
  * Pregnant or breastfeeding.
  * Known hypersensitivity to perflutren (contained in Definity

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 17 Healthy controls and 17 participants with T1D
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Myocardial Microvascular Perfusion (measured by contrast-enhanced ultrasound) | baseline and 2 hours after a meal
  Measurement of change in myocardial microvascular perfusion

SECONDARY OUTCOMES:
Skeletal Muscle Microvascular Perfusion (measured by contrast-enhanced ultrasound) | baseline and 2 hours after a meal
  Measurement of change in microvascular perfusion of skeletal muscle
Flow Mediated Dilation | baseline and 2 hours after a meal
  Vascular measure of change in conduit artery stiffness
Pulse Wave Velocity ( PWV) | baseline and 2 hours after a meal
  Measurement of change in central artery stiffness
Tumor Necrosis Factor-Alpha (TNF-alpha) | baseline and 2 hours after a meal
  Inflammatory biomarker (plasma sample) specific specific to patients with type 1 diabetes
Interleukin 6 (IL-6) | baseline and 2 hours after a meal
  Inflammatory biomarker (plasma sample) specific specific to patients with type 1 diabetes
high sensitivity C-reactive protein (hsCRP) | baseline and 2 hours after a meal
  Inflammatory biomarker (plasma sample) specific specific to patients with type 1 diabetes
Intercellular Adhesion Molecule 1 (ICAM-1) | baseline and 2 hours after a meal
  Biomarker (plasma sample) of endothelial dysfunction
E-selectin | baseline and 2 hours after a meal
  Biomarker (plasma sample) of endothelial dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: William Horton, MD, Principal Investigator — University of Virginia, Department of Endocrinology; Zhenqi Liu, MD, Study Chair — University of Virginia, Department of Endocrinology
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Lind M, Svensson AM, Kosiborod M, Gudbjornsdottir S, Pivodic A, Wedel H, Dahlqvist S, Clements M, Rosengren A. Glycemic control and excess mortality in type 1 diabetes. N Engl J Med. 2014 Nov 20;371(21):1972-82. doi: 10.1056/NEJMoa1408214. PMID 25409370
- [Background] Lee AK, Warren B, Lee CJ, McEvoy JW, Matsushita K, Huang ES, Sharrett AR, Coresh J, Selvin E. The Association of Severe Hypoglycemia With Incident Cardiovascular Events and Mortality in Adults With Type 2 Diabetes. Diabetes Care. 2018 Jan;41(1):104-111. doi: 10.2337/dc17-1669. Epub 2017 Nov 10. PMID 29127240
- [Background] Goto A, Goto M, Terauchi Y, Yamaguchi N, Noda M. Association Between Severe Hypoglycemia and Cardiovascular Disease Risk in Japanese Patients With Type 2 Diabetes. J Am Heart Assoc. 2016 Mar 9;5(3):e002875. doi: 10.1161/JAHA.115.002875. PMID 26961698
- [Background] Aryangat AV, Gerich JE. Type 2 diabetes: postprandial hyperglycemia and increased cardiovascular risk. Vasc Health Risk Manag. 2010 Mar 24;6:145-55. doi: 10.2147/vhrm.s8216. PMID 20448799
- [Background] Ceriello A, Hanefeld M, Leiter L, Monnier L, Moses A, Owens D, Tajima N, Tuomilehto J. Postprandial glucose regulation and diabetic complications. Arch Intern Med. 2004 Oct 25;164(19):2090-5. doi: 10.1001/archinte.164.19.2090. PMID 15505121
- [Background] Cavalot F, Petrelli A, Traversa M, Bonomo K, Fiora E, Conti M, Anfossi G, Costa G, Trovati M. Postprandial blood glucose is a stronger predictor of cardiovascular events than fasting blood glucose in type 2 diabetes mellitus, particularly in women: lessons from the San Luigi Gonzaga Diabetes Study. J Clin Endocrinol Metab. 2006 Mar;91(3):813-9. doi: 10.1210/jc.2005-1005. Epub 2005 Dec 13. PMID 16352690
- [Background] Livingstone SJ, Looker HC, Hothersall EJ, Wild SH, Lindsay RS, Chalmers J, Cleland S, Leese GP, McKnight J, Morris AD, Pearson DW, Peden NR, Petrie JR, Philip S, Sattar N, Sullivan F, Colhoun HM. Risk of cardiovascular disease and total mortality in adults with type 1 diabetes: Scottish registry linkage study. PLoS Med. 2012;9(10):e1001321. doi: 10.1371/journal.pmed.1001321. Epub 2012 Oct 2. PMID 23055834
- [Background] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Background] Currie CJ, Peters JR, Tynan A, Evans M, Heine RJ, Bracco OL, Zagar T, Poole CD. Survival as a function of HbA(1c) in people with type 2 diabetes: a retrospective cohort study. Lancet. 2010 Feb 6;375(9713):481-9. doi: 10.1016/S0140-6736(09)61969-3. Epub 2010 Jan 26. PMID 20110121
- [Background] Saisho Y. Glycemic variability and oxidative stress: a link between diabetes and cardiovascular disease? Int J Mol Sci. 2014 Oct 13;15(10):18381-406. doi: 10.3390/ijms151018381. PMID 25314300
- [Background] Risso A, Mercuri F, Quagliaro L, Damante G, Ceriello A. Intermittent high glucose enhances apoptosis in human umbilical vein endothelial cells in culture. Am J Physiol Endocrinol Metab. 2001 Nov;281(5):E924-30. doi: 10.1152/ajpendo.2001.281.5.E924. PMID 11595647
- [Background] Quagliaro L, Piconi L, Assaloni R, Martinelli L, Motz E, Ceriello A. Intermittent high glucose enhances apoptosis related to oxidative stress in human umbilical vein endothelial cells: the role of protein kinase C and NAD(P)H-oxidase activation. Diabetes. 2003 Nov;52(11):2795-804. doi: 10.2337/diabetes.52.11.2795. PMID 14578299
- [Background] Piconi L, Quagliaro L, Assaloni R, Da Ros R, Maier A, Zuodar G, Ceriello A. Constant and intermittent high glucose enhances endothelial cell apoptosis through mitochondrial superoxide overproduction. Diabetes Metab Res Rev. 2006 May-Jun;22(3):198-203. doi: 10.1002/dmrr.613. PMID 16453381
- [Background] Horvath EM, Benko R, Kiss L, Muranyi M, Pek T, Fekete K, Barany T, Somlai A, Csordas A, Szabo C. Rapid 'glycaemic swings' induce nitrosative stress, activate poly(ADP-ribose) polymerase and impair endothelial function in a rat model of diabetes mellitus. Diabetologia. 2009 May;52(5):952-61. doi: 10.1007/s00125-009-1304-0. Epub 2009 Mar 5. PMID 19263033
- [Background] Ceriello A, Esposito K, Piconi L, Ihnat MA, Thorpe JE, Testa R, Boemi M, Giugliano D. Oscillating glucose is more deleterious to endothelial function and oxidative stress than mean glucose in normal and type 2 diabetic patients. Diabetes. 2008 May;57(5):1349-54. doi: 10.2337/db08-0063. Epub 2008 Feb 25. PMID 18299315
- [Background] Monnier L, Mas E, Ginet C, Michel F, Villon L, Cristol JP, Colette C. Activation of oxidative stress by acute glucose fluctuations compared with sustained chronic hyperglycemia in patients with type 2 diabetes. JAMA. 2006 Apr 12;295(14):1681-7. doi: 10.1001/jama.295.14.1681. PMID 16609090
- [Background] Tang X, Li S, Wang Y, Wang M, Yin Q, Mu P, Lin S, Qian X, Ye X, Chen Y. Glycemic variability evaluated by continuous glucose monitoring system is associated with the 10-y cardiovascular risk of diabetic patients with well-controlled HbA1c. Clin Chim Acta. 2016 Oct 1;461:146-50. doi: 10.1016/j.cca.2016.08.004. Epub 2016 Aug 5. PMID 27502250
- [Background] Ghouse J, Skov MW, Kanters JK, Lind B, Isaksen JL, Blanche P, Haunso S, Kober L, Svendsen JH, Olesen MS, Holst AG, Gerds TA, Nielsen JB. Visit-to-Visit Variability of Hemoglobin A1c in People Without Diabetes and Risk of Major Adverse Cardiovascular Events and All-Cause Mortality. Diabetes Care. 2019 Jan;42(1):134-141. doi: 10.2337/dc18-1396. Epub 2018 Oct 23. PMID 30352898
- [Background] Su G, Mi SH, Tao H, Li Z, Yang HX, Zheng H, Zhou Y, Tian L. Impact of admission glycemic variability, glucose, and glycosylated hemoglobin on major adverse cardiac events after acute myocardial infarction. Diabetes Care. 2013 Apr;36(4):1026-32. doi: 10.2337/dc12-0925. Epub 2013 Jan 24. PMID 23349547
- [Background] Waden J, Forsblom C, Thorn LM, Gordin D, Saraheimo M, Groop PH; Finnish Diabetic Nephropathy Study Group. A1C variability predicts incident cardiovascular events, microalbuminuria, and overt diabetic nephropathy in patients with type 1 diabetes. Diabetes. 2009 Nov;58(11):2649-55. doi: 10.2337/db09-0693. Epub 2009 Aug 3. PMID 19651819
- [Background] Snell-Bergeon JK, Roman R, Rodbard D, Garg S, Maahs DM, Schauer IE, Bergman BC, Kinney GL, Rewers M. Glycaemic variability is associated with coronary artery calcium in men with Type 1 diabetes: the Coronary Artery Calcification in Type 1 Diabetes study. Diabet Med. 2010 Dec;27(12):1436-42. doi: 10.1111/j.1464-5491.2010.03127.x. PMID 21059097
- [Background] Sundell J, Knuuti J. Insulin and myocardial blood flow. Cardiovasc Res. 2003 Feb;57(2):312-9. doi: 10.1016/s0008-6363(02)00718-6. PMID 12566104
- [Background] Coggins M, Lindner J, Rattigan S, Jahn L, Fasy E, Kaul S, Barrett E. Physiologic hyperinsulinemia enhances human skeletal muscle perfusion by capillary recruitment. Diabetes. 2001 Dec;50(12):2682-90. doi: 10.2337/diabetes.50.12.2682. PMID 11723050
- [Background] Vincent MA, Dawson D, Clark AD, Lindner JR, Rattigan S, Clark MG, Barrett EJ. Skeletal muscle microvascular recruitment by physiological hyperinsulinemia precedes increases in total blood flow. Diabetes. 2002 Jan;51(1):42-8. doi: 10.2337/diabetes.51.1.42. PMID 11756321
- [Background] de Ferranti SD, de Boer IH, Fonseca V, Fox CS, Golden SH, Lavie CJ, Magge SN, Marx N, McGuire DK, Orchard TJ, Zinman B, Eckel RH. Type 1 diabetes mellitus and cardiovascular disease: a scientific statement from the American Heart Association and American Diabetes Association. Diabetes Care. 2014 Oct;37(10):2843-63. doi: 10.2337/dc14-1720. Epub 2014 Aug 11. No abstract available. PMID 25114297
- [Background] Martin-Timon I, Sevillano-Collantes C, Segura-Galindo A, Del Canizo-Gomez FJ. Type 2 diabetes and cardiovascular disease: Have all risk factors the same strength? World J Diabetes. 2014 Aug 15;5(4):444-70. doi: 10.4239/wjd.v5.i4.444. PMID 25126392
- [Background] Priya G, Kalra S. A Review of Insulin Resistance in Type 1 Diabetes: Is There a Place for Adjunctive Metformin? Diabetes Ther. 2018 Feb;9(1):349-361. doi: 10.1007/s13300-017-0333-9. Epub 2017 Nov 14. PMID 29139080
- [Background] Alessa T, Szeto A, Chacra W, Mendez A, Goldberg RB. High HDL-C prevalence is common in type 1 diabetes and increases with age but is lower in Hispanic individuals. J Diabetes Complications. 2015 Jan-Feb;29(1):105-7. doi: 10.1016/j.jdiacomp.2014.08.011. Epub 2014 Sep 6. PMID 25441221
- [Background] Norgaard K, Feldt-Rasmussen B, Borch-Johnsen K, Saelan H, Deckert T. Prevalence of hypertension in type 1 (insulin-dependent) diabetes mellitus. Diabetologia. 1990 Jul;33(7):407-10. doi: 10.1007/BF00404089. PMID 2401396
- [Background] Corbin KD, Driscoll KA, Pratley RE, Smith SR, Maahs DM, Mayer-Davis EJ; Advancing Care for Type 1 Diabetes and Obesity Network (ACT1ON). Obesity in Type 1 Diabetes: Pathophysiology, Clinical Impact, and Mechanisms. Endocr Rev. 2018 Oct 1;39(5):629-663. doi: 10.1210/er.2017-00191. PMID 30060120
- [Background] Gorst C, Kwok CS, Aslam S, Buchan I, Kontopantelis E, Myint PK, Heatlie G, Loke Y, Rutter MK, Mamas MA. Long-term Glycemic Variability and Risk of Adverse Outcomes: A Systematic Review and Meta-analysis. Diabetes Care. 2015 Dec;38(12):2354-69. doi: 10.2337/dc15-1188. PMID 26604281
- [Background] Bonke FC, Donnachie E, Schneider A, Mehring M. Association of the average rate of change in HbA1c with severe adverse events: a longitudinal evaluation of audit data from the Bavarian Disease Management Program for patients with type 2 diabetes mellitus. Diabetologia. 2016 Feb;59(2):286-93. doi: 10.1007/s00125-015-3797-z. Epub 2015 Oct 30. PMID 26518684
- [Background] Wan EY, Fung CS, Fong DY, Lam CL. Association of variability in hemoglobin A1c with cardiovascular diseases and mortality in Chinese patients with type 2 diabetes mellitus - A retrospective population-based cohort study. J Diabetes Complications. 2016 Sep-Oct;30(7):1240-7. doi: 10.1016/j.jdiacomp.2016.05.024. Epub 2016 May 31. PMID 27318537
- [Background] Lee CL, Sheu WH, Lee IT, Lin SY, Liang WM, Wang JS, Li YF. Trajectories of fasting plasma glucose variability and mortality in type 2 diabetes. Diabetes Metab. 2018 Mar;44(2):121-128. doi: 10.1016/j.diabet.2017.09.001. Epub 2017 Oct 9. PMID 29032950
- [Background] Wightman SS, Sainsbury CAR, Jones GC. Visit-to-visit HbA1c variability and systolic blood pressure (SBP) variability are significantly and additively associated with mortality in individuals with type 1 diabetes: An observational study. Diabetes Obes Metab. 2018 Apr;20(4):1014-1017. doi: 10.1111/dom.13193. Epub 2018 Jan 18. PMID 29266630
- [Background] Gerbaud E, Darier R, Montaudon M, Beauvieux MC, Coffin-Boutreux C, Coste P, Douard H, Ouattara A, Catargi B. Glycemic Variability Is a Powerful Independent Predictive Factor of Midterm Major Adverse Cardiac Events in Patients With Diabetes With Acute Coronary Syndrome. Diabetes Care. 2019 Apr;42(4):674-681. doi: 10.2337/dc18-2047. Epub 2019 Feb 6. PMID 30728222
- [Background] Vincent MA, Clerk LH, Lindner JR, Price WJ, Jahn LA, Leong-Poi H, Barrett EJ. Mixed meal and light exercise each recruit muscle capillaries in healthy humans. Am J Physiol Endocrinol Metab. 2006 Jun;290(6):E1191-7. doi: 10.1152/ajpendo.00497.2005. PMID 16682488
- [Background] Chai W, Liu J, Jahn LA, Fowler DE, Barrett EJ, Liu Z. Salsalate attenuates free fatty acid-induced microvascular and metabolic insulin resistance in humans. Diabetes Care. 2011 Jul;34(7):1634-8. doi: 10.2337/dc10-2345. Epub 2011 May 26. PMID 21617098
- [Background] Subaran SC, Sauder MA, Chai W, Jahn LA, Fowler DE, Aylor KW, Basu A, Liu Z. GLP-1 at physiological concentrations recruits skeletal and cardiac muscle microvasculature in healthy humans. Clin Sci (Lond). 2014 Aug;127(3):163-70. doi: 10.1042/CS20130708. PMID 24552454
- [Background] Jahn LA, Hartline L, Rao N, Logan B, Kim JJ, Aylor K, Gan LM, Westergren HU, Barrett EJ. Insulin Enhances Endothelial Function Throughout the Arterial Tree in Healthy But Not Metabolic Syndrome Subjects. J Clin Endocrinol Metab. 2016 Mar;101(3):1198-206. doi: 10.1210/jc.2015-3293. Epub 2016 Jan 12. PMID 26756115
- [Background] Liu J, Jahn LA, Fowler DE, Barrett EJ, Cao W, Liu Z. Free fatty acids induce insulin resistance in both cardiac and skeletal muscle microvasculature in humans. J Clin Endocrinol Metab. 2011 Feb;96(2):438-46. doi: 10.1210/jc.2010-1174. Epub 2010 Nov 3. PMID 21047922
- [Background] Zorach B, Shaw PW, Bourque J, Kuruvilla S, Balfour PC Jr, Yang Y, Mathew R, Pan J, Gonzalez JA, Taylor AM, Meyer CH, Epstein FH, Kramer CM, Salerno M. Quantitative cardiovascular magnetic resonance perfusion imaging identifies reduced flow reserve in microvascular coronary artery disease. J Cardiovasc Magn Reson. 2018 Feb 22;20(1):14. doi: 10.1186/s12968-018-0435-1. PMID 29471856
- [Background] Jamiolkowska M, Jamiolkowska I, Luczynski W, Tolwinska J, Bossowski A, Glowinska Olszewska B. Impact of Real-Time Continuous Glucose Monitoring Use on Glucose Variability and Endothelial Function in Adolescents with Type 1 Diabetes: New Technology--New Possibility to Decrease Cardiovascular Risk? J Diabetes Res. 2016;2016:4385312. doi: 10.1155/2016/4385312. Epub 2015 Nov 16. PMID 26649320
- [Background] Rana O, Byrne CD, Kerr D, Coppini DV, Zouwail S, Senior R, Begley J, Walker JJ, Greaves K. Acute hypoglycemia decreases myocardial blood flow reserve in patients with type 1 diabetes mellitus and in healthy humans. Circulation. 2011 Oct 4;124(14):1548-56. doi: 10.1161/CIRCULATIONAHA.110.992297. Epub 2011 Sep 12. PMID 21911786
- [Background] Abdelmoneim SS, Hagen ME, Mendrick E, Pattan V, Wong B, Norby B, Roberson T, Szydel T, Basu R, Basu A, Mulvagh SL. Acute hyperglycemia reduces myocardial blood flow reserve and the magnitude of reduction is associated with insulin resistance: a study in nondiabetic humans using contrast echocardiography. Heart Vessels. 2013 Nov;28(6):757-68. doi: 10.1007/s00380-012-0305-y. Epub 2012 Nov 23. PMID 23180239
- [Background] Davis SN, Duckworth W, Emanuele N, Hayward RA, Wiitala WL, Thottapurathu L, Reda DJ, Reaven PD; Investigators of the Veterans Affairs Diabetes Trial. Effects of Severe Hypoglycemia on Cardiovascular Outcomes and Death in the Veterans Affairs Diabetes Trial. Diabetes Care. 2019 Jan;42(1):157-163. doi: 10.2337/dc18-1144. Epub 2018 Nov 19. PMID 30455335
- [Background] Zinman B, Marso SP, Christiansen E, Calanna S, Rasmussen S, Buse JB; LEADER Publication Committee on behalf of the LEADER Trial Investigators. Hypoglycemia, Cardiovascular Outcomes, and Death: The LEADER Experience. Diabetes Care. 2018 Aug;41(8):1783-1791. doi: 10.2337/dc17-2677. Epub 2018 Jun 14. PMID 29903847
- [Background] Ceriello A. The emerging role of post-prandial hyperglycaemic spikes in the pathogenesis of diabetic complications. Diabet Med. 1998 Mar;15(3):188-93. doi: 10.1002/(SICI)1096-9136(199803)15:33.0.CO;2-V. No abstract available. PMID 9545118
- [Background] Glucose tolerance and mortality: comparison of WHO and American Diabetes Association diagnostic criteria. The DECODE study group. European Diabetes Epidemiology Group. Diabetes Epidemiology: Collaborative analysis Of Diagnostic criteria in Europe. Lancet. 1999 Aug 21;354(9179):617-21. PMID 10466661
- [Background] Strojek K, Raz I, Jermendy G, Gitt AK, Liu R, Zhang Q, Jacober SJ, Milicevic Z. Factors Associated With Cardiovascular Events in Patients With Type 2 Diabetes and Acute Myocardial Infarction. J Clin Endocrinol Metab. 2016 Jan;101(1):243-53. doi: 10.1210/jc.2015-1962. Epub 2015 Nov 23. PMID 26595100
- [Background] Scognamiglio R, Negut C, De Kreutzenberg SV, Tiengo A, Avogaro A. Postprandial myocardial perfusion in healthy subjects and in type 2 diabetic patients. Circulation. 2005 Jul 12;112(2):179-84. doi: 10.1161/CIRCULATIONAHA.104.495127. Epub 2005 Jul 5. PMID 15998667
- [Background] Scognamiglio R, Negut C, de Kreutzenberg SV, Tiengo A, Avogaro A. Effects of different insulin regimes on postprandial myocardial perfusion defects in type 2 diabetic patients. Diabetes Care. 2006 Jan;29(1):95-100. PMID 16373903
- [Background] Haas AV, Rosner BA, Kwong RY, Rao AD, Garg R, Di Carli MF, Adler GK. Sex Differences in Coronary Microvascular Function in Individuals With Type 2 Diabetes. Diabetes. 2019 Mar;68(3):631-636. doi: 10.2337/db18-0650. Epub 2018 Nov 8. PMID 30409780
- [Background] Bagi Z, Broskova Z, Feher A. Obesity and coronary microvascular disease - implications for adipose tissue-mediated remote inflammatory response. Curr Vasc Pharmacol. 2014 May;12(3):453-61. doi: 10.2174/1570161112666140423221843. PMID 24846234
- [Background] Larghat AM, Swoboda PP, Biglands JD, Kearney MT, Greenwood JP, Plein S. The microvascular effects of insulin resistance and diabetes on cardiac structure, function, and perfusion: a cardiovascular magnetic resonance study. Eur Heart J Cardiovasc Imaging. 2014 Dec;15(12):1368-76. doi: 10.1093/ehjci/jeu142. Epub 2014 Aug 12. PMID 25117473
- [Background] Barletta G, Del Bene MR. Myocardial perfusion echocardiography and coronary microvascular dysfunction. World J Cardiol. 2015 Dec 26;7(12):861-74. doi: 10.4330/wjc.v7.i12.861. PMID 26730291
- [Background] Kuruvilla S, Janardhanan R, Antkowiak P, Keeley EC, Adenaw N, Brooks J, Epstein FH, Kramer CM, Salerno M. Increased extracellular volume and altered mechanics are associated with LVH in hypertensive heart disease, not hypertension alone. JACC Cardiovasc Imaging. 2015 Feb;8(2):172-80. doi: 10.1016/j.jcmg.2014.09.020. Epub 2015 Jan 7. PMID 25577446
- [Background] Monnier L, Colette C, Owens DR. Glycemic variability: the third component of the dysglycemia in diabetes. Is it important? How to measure it? J Diabetes Sci Technol. 2008 Nov;2(6):1094-100. doi: 10.1177/193229680800200618. PMID 19885298
- [Background] Miller RG, Costacou T, Orchard TJ. Risk Factor Modeling for Cardiovascular Disease in Type 1 Diabetes in the Pittsburgh Epidemiology of Diabetes Complications (EDC) Study: A Comparison With the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Study (DCCT/EDIC). Diabetes. 2019 Feb;68(2):409-419. doi: 10.2337/db18-0515. Epub 2018 Nov 8. PMID 30409781
- [Background] Tam CS, Xie W, Johnson WD, Cefalu WT, Redman LM, Ravussin E. Defining insulin resistance from hyperinsulinemic-euglycemic clamps. Diabetes Care. 2012 Jul;35(7):1605-10. doi: 10.2337/dc11-2339. Epub 2012 Apr 17. PMID 22511259
- [Background] Chan A, Barrett EJ, Anderson SM, Kovatchev BP, Breton MD. Muscle microvascular recruitment predicts insulin sensitivity in middle-aged patients with type 1 diabetes mellitus. Diabetologia. 2012 Mar;55(3):729-36. doi: 10.1007/s00125-011-2402-3. Epub 2011 Dec 14. PMID 22167126
- [Background] Breton MD, Patek SD, Lv D, Schertz E, Robic J, Pinnata J, Kollar L, Barnett C, Wakeman C, Oliveri M, Fabris C, Chernavvsky D, Kovatchev BP, Anderson SM. Continuous Glucose Monitoring and Insulin Informed Advisory System with Automated Titration and Dosing of Insulin Reduces Glucose Variability in Type 1 Diabetes Mellitus. Diabetes Technol Ther. 2018 Aug;20(8):531-540. doi: 10.1089/dia.2018.0079. Epub 2018 Jul 6. PMID 29979618
- [Background] Monnier L, Colette C, Wojtusciszyn A, Dejager S, Renard E, Molinari N, Owens DR. Toward Defining the Threshold Between Low and High Glucose Variability in Diabetes. Diabetes Care. 2017 Jul;40(7):832-838. doi: 10.2337/dc16-1769. Epub 2016 Dec 30. PMID 28039172
- [Background] Kovatchev B, Cobelli C. Glucose Variability: Timing, Risk Analysis, and Relationship to Hypoglycemia in Diabetes. Diabetes Care. 2016 Apr;39(4):502-10. doi: 10.2337/dc15-2035. PMID 27208366
- [Background] Danne T, Nimri R, Battelino T, Bergenstal RM, Close KL, DeVries JH, Garg S, Heinemann L, Hirsch I, Amiel SA, Beck R, Bosi E, Buckingham B, Cobelli C, Dassau E, Doyle FJ 3rd, Heller S, Hovorka R, Jia W, Jones T, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Maahs D, Murphy HR, Norgaard K, Parkin CG, Renard E, Saboo B, Scharf M, Tamborlane WV, Weinzimer SA, Phillip M. International Consensus on Use of Continuous Glucose Monitoring. Diabetes Care. 2017 Dec;40(12):1631-1640. doi: 10.2337/dc17-1600. PMID 29162583
- [Background] Ohkuma T, Komorita Y, Peters SAE, Woodward M. Diabetes as a risk factor for heart failure in women and men: a systematic review and meta-analysis of 47 cohorts including 12 million individuals. Diabetologia. 2019 Sep;62(9):1550-1560. doi: 10.1007/s00125-019-4926-x. Epub 2019 Jul 18. PMID 31317230
- [Background] Lind M, Bounias I, Olsson M, Gudbjornsdottir S, Svensson AM, Rosengren A. Glycaemic control and incidence of heart failure in 20,985 patients with type 1 diabetes: an observational study. Lancet. 2011 Jul 9;378(9786):140-6. doi: 10.1016/S0140-6736(11)60471-6. Epub 2011 Jun 24. PMID 21705065
- [Background] Tromp J, Lim SL, Tay WT, Teng TK, Chandramouli C, Ouwerkerk W, Wander GS, Sawhney JPS, Yap J, MacDonald MR, Ling LH, Sattar N, McMurray JJV, Richards AM, Anand I, Lam CSP; ASIAN-HF Investigators. Microvascular Disease in Patients With Diabetes With Heart Failure and Reduced Ejection Versus Preserved Ejection Fraction. Diabetes Care. 2019 Sep;42(9):1792-1799. doi: 10.2337/dc18-2515. Epub 2019 Jul 10. PMID 31292141
- [Background] Su MY, Lin LY, Tseng YH, Chang CC, Wu CK, Lin JL, Tseng WY. CMR-verified diffuse myocardial fibrosis is associated with diastolic dysfunction in HFpEF. JACC Cardiovasc Imaging. 2014 Oct;7(10):991-7. doi: 10.1016/j.jcmg.2014.04.022. Epub 2014 Sep 17. PMID 25240451
- [Background] Ng AC, Auger D, Delgado V, van Elderen SG, Bertini M, Siebelink HM, van der Geest RJ, Bonetti C, van der Velde ET, de Roos A, Smit JW, Leung DY, Bax JJ, Lamb HJ. Association between diffuse myocardial fibrosis by cardiac magnetic resonance contrast-enhanced T(1) mapping and subclinical myocardial dysfunction in diabetic patients: a pilot study. Circ Cardiovasc Imaging. 2012 Jan;5(1):51-9. doi: 10.1161/CIRCIMAGING.111.965608. Epub 2011 Dec 1. PMID 22135399
- [Background] Mavrogeni S, Bratis K, Gavra P, Fousteris E, Markussis V, Kolovou G, van Wijk K, Hautemann D, Reiber JH, Melidonis A. Stress cardiac magnetic resonance reveals myocardial perfusion impairment in asymptomatic diabetes mellitus type I, missed by the routine non-invasive evaluation. Int J Cardiol. 2013 Sep 10;167(6):e167-9. doi: 10.1016/j.ijcard.2013.04.170. Epub 2013 May 9. No abstract available. PMID 23664053
- [Background] Turkbey EB, Backlund JY, Genuth S, Jain A, Miao C, Cleary PA, Lachin JM, Nathan DM, van der Geest RJ, Soliman EZ, Liu CY, Lima JA, Bluemke DA; DCCT/EDIC Research Group. Myocardial structure, function, and scar in patients with type 1 diabetes mellitus. Circulation. 2011 Oct 18;124(16):1737-46. doi: 10.1161/CIRCULATIONAHA.111.022327. Epub 2011 Sep 26. PMID 21947298